CLINICAL TRIAL: NCT05717725
Title: Pulsed-field Ablation Versus Sham Ablation to Treat Atrial Fibrillation
Brief Title: Pulsed-field Ablation Vs. Sham Ablation to Treat AF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Na Homolce Hospital (Other); Nemocnice AGEL Trinec-Podlesi a.s. (Other); Neuron Medical s.r.o. (Unknown)
Responsible Party: Principal Investigator, Pavel Osmancik, head of the dept. of cardiac arrhythmias, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PFA SHAM
Record Dates: First submitted 2022-10-31; First posted 2023-02-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; pulsed-field ablation; quality of life
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to pulsed-field ablation or sham procedure.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed-field ablation arm (Active Comparator): Patients will undergo catheter ablation using for atrial fibrillation using pulsed-field energy
  Interventions: Procedure: Pulsed-field ablation
- Sham procedure arm (Sham Comparator): Patients will receive sham procedure (no ablation)
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Pulsed-field ablation — Patients will receive catheter ablation, i.e. pulmonary vein isolation by means of pulsed-field energy
  Arms: Pulsed-field ablation arm
Procedure: Sham procedure — Patients will receive sham procedure, no ablation.
  Arms: Sham procedure arm

SUMMARY:
The study is planned as a single-blind, multicenter, prospective, randomized study. Sixty sbjects will be randomized 1:1 to either: (i) EP study + PFA, or (ii) EP study + Sham ablation control.

After informed consent is obtained, an implantable loop recorder (ILR) will be implanted within seven days, and an EP study will be scheduled for 30±5 days after ILR implantation.

Patients in both groups will first undergo an EP study to rule out a concealed AV bypass tract and supraventricular tachycardia (SVT). Patients will not be randomized if SVT or concealed AV bypass tract is found during the EP study. Once an SVT or bypass tract is excluded, randomization will be performed. Patients randomized to Ablation will undergo PVI using the commercially-available pentaspline PFA catheter (Farawave, Farapulse-BSCI Inc). Patients randomized to the Sham-ablation Control group will simply undergo approximately 20-30 min of anesthesia with propofol and benzodiazepines in a similar manner as patients in the ablation arm.

Primary endpoints will be assessed six months after the procedure.

ECGs will be monitored using implantable ECG monitors (ILR) in all patients. There will be two co-primary endpoints (assessed at six months or at cross-over if Early Exit):

1. Freedom from recurrent AF/AT/AFL (post 2-month blanking), assessed as time-to first recurrence;
2. Quality of life according to Atrial Fibrillation Effect on QualiTy of life (AFEQT) score at 6 months (or at cross-over if Early Exit).

DETAILED DESCRIPTION:
PURPOSE The purpose of PFA-Sham is to determine the relative efficacy of catheter ablation for symptomatic paroxysmal/persistent AF, when compared against a sham-ablation control procedure. This is a prospective, multi-center, single-blind, randomized trial.

There are two co-primary hypotheses. First, we hypothesize that patients in the catheter ablation group will experience greater freedom from recurrent AF/AT/AFL at 6 months post-procedure. There will be a two-month post-procedure blanking period in both groups. Freedom from AF/AT/AFL will be assessed as time to first recurrence (or to cross-over if earlier).

Second, compared with those in the sham-ablation control group, patients in the catheter ablation group will report higher quality of life as measured by the Atrial Fibrillation Effect on QualiTy of life (AFEQT) score, at 6 months post-procedure (or at cross-over if Early Exit).

METHODS The study will be a single-blind, multicenter, prospective, randomized control study. Subjects will be randomized 1:1 to either: (i) EP study + PFA, or (ii) EP study + Sham ablation control.

After informed consent is obtained, an implantable loop recorder (ILR) will be implanted within seven days, and an EP study will be scheduled for 30±5 days after ILR implantation.

Patients in both groups will first undergo an EP study to rule out a concealed AV bypass tract and supraventricular tachycardia (SVT), and catheter ablation of this substrate if present. Patients will not be randomized if SVT or concealed AV bypass tract is found during the EP study.

Once an SVT or bypass tract is excluded, randomization will be performed. Patients randomized to Ablation will undergo PVI using the commercially-available pentaspline PFA catheter (Farawave, Farapulse-BSCI Inc). Patients randomized to the Sham-ablation Control group will undergo approximately 20-30 min of anesthesia with propofol and benzodiazepines in a similar manner as patients in the ablation arm.

INCLUSION CRITERIA

1. Age >18 years
2. Paroxysmal or Persistent Atrial Fibrillation (but not long-standing Persistent AF)
3. Screening (qualifying) AFEQT score ≤ 50

AF symptoms will be assessed using the AFEQT questionnaire during screening. AFEQT is a 20-item questionnaire, and provides a 4-item Symptoms score, an 8-item Daily Activities score, a 6-item Treatment Concerns score, and a 2-item Treatment Satisfaction scale. Overall and subscale scores range from 0 to 100. A score of 0 corresponds to complete disability, while a score of 100 describes the highest level of QOL.In the study, screening (qualifying) AFEQT score has to be less than 50.

EXCLUSION CRITERIA

1. Any prior AF ablation procedure (or left atrial ablation procedure)
2. Untreated other arrhythmias (e.g. atrial flutter, SVT, VT, frequent PVCs);
3. Long-standing Persistent AF episodes (any continuous episodes lasting > 1 year);
4. Permanent AF;
5. No ECG evidence of AF episode >30 seconds in the 6 months prior to randomization;
6. LA size > 55 mm;
7. Hypertrophic cardiomyopathy;
8. Valve disease (any aortic stenosis, moderate or severe mitral regurgitation);
9. Left ventricular ejection fraction ≤ 35% according to echocardiogram within 6 months of randomization;
10. Moderate or severe pulmonary hypertension
11. History of tachycardia-induced cardiomyopathy;
12. Symptomatic coronary artery disease;
13. Pregnancy;
14. Presence of an artificial valve;
15. Life expectancy less than two years;
16. Known medical condition or contraindication causing potential complications for interventional procedures or follow up

ENROLLMENT AND ILR IMPLANT

Data will be gathered including the following:

* Demographics including gender, height and weight
* Pertinent medical and cardiovascular history, CHA2DS2-VASc
* AAD and anticoagulation medication history
* 12-lead ECG
* TTE within 6 months
* The Atrial Fibrillation Effect on QualiTy-of-Life Questionnaire (AFEQT) quality of life assessment at enrollment

EP STUDY, AFEQT and HADS Before randomization, all patients will undergo an electrophysiology (EP) study. An EP study will be scheduled at 30 days after ILR implantation. Within 1 day of the procedure, all patients will have assessment of the baseline AFEQT and Hospital Anxiety and Depression Scale (HADS), and atrial arrhythmia burden by interrogation of their ILR. (The HADS scale is a 14-item instrument that evaluates symptoms of anxiety and depression in medical populations, on a 4-point scale from 0 to 3. These data (baseline AFEQT, baseline HADS, and ILR interogation) will constitute baseline measurements for the purpose of endpoint estimation.

The EP study will be done using standard techniques; two EP catheters will be inserted via one femoral vein. Femoral access should be performed with ultrasound guidance. One catheter will be inserted in the coronary sinus, the other at the His bundle area. SVT and concealed accessory pathway (AP) will be excluded using standard EP protocols (retrograde ventricular pacing to exclude concealed AP, programmed atrial stimulation to exclude dual AV node physiology, and AV nodal reentry initiation). If concealed AP or inducible AVNRT is present, the arrhythmia will be targeted, but the patient cannot be randomized. These patients will be further monitored in the outpatient clinic as NON-randomized patients. These patients that sign consent but undergo SVT ablation do not count to the 60-patient enrollment goal.

If SVT or concealed AP are excluded, patients will be randomized to the catheter ablation group (CA) or Control Sham group) in a 1:1 ratio.

Group 1: catheter ablation; or Group 2: sham ablation (control group).

RANDOMIZATION will be done using web-based randomization software at the end of the EP procedure. The software will be designed to account for gender and the type of AF (paroxysmal/non-paroxysmal), with the goal of having comparable groups regarding the type of AF. The randomization process will be done outside all participating centers using an electronic web-based CRF; therefore, it will be independent of study subjects and site personnel. No physicia at later out-patient controls will have information on the arm in which the patient was randomized.

TREATMENTS Ablation Arm: after the EP study, patients will undergo pulmonary vein isolation (PVI) using a PFA catheter (Farawave; Farapulse-BSCI Inc.). The same vascular (venous) access used in the EP study will be used for catheter insertion. PFA energy will be applied according to the recommendation of the manufactureur. At the end of the procedure, a single figure-of-eight suture can be placed to achieve hemostasis. The whole procedure will be done under analgosedation (propofol, benzodiazepines, ketamine, opioids) and with the guidance of an anesthesiologist, or as per the center standard of care.

Control arm: after the EP study, patients should undergo approximately 20-30 min of anesthesia with propofol and benzodiazepines in a similar manner as patients in the ablation arm. An anesthesiologist will guide the analgosedation, or as per the center standard of care. At the end of the procedure, a figure-of-eight suture will be placed.

After the procedure, patients will be monitored in the hospital, followed by a TTE to rule out a pericardial effusion. Patients will be discharged the day after the procedure.

Before hospital discharge (ideally the day after the procedure), patients will complete the baseline Blinding Questionnaire.

In-person assessments at months 2, 3, 6 and 12 months post-procedure

* ECG
* Adverse events
* AAD and anticoagulation medication use
* Recurrent arrhythmia, cardioversions, ablations, hospital admissions
* AF/AT/AFL burden assessment at 6 months and 12 months only (ILR interrogation to core lab)
* The Atrial Fibrillation Effect on QualiTy-of-Life Questionnaire (AFEQT) quality of life assessment
* Hospital Anxiety and Depression Scale (HADS) score (at 2 and 6 months only)
* Blinding Questionnaire (at 2 and 6 months only)

Assessments at months 1, 4, 5, 9 post-procedure

These will be performed by phone, and will include the following elements:

* Adverse events
* AAD and anticoagulation medication use
* Recurrent arrhythmia, cardioversions, ablations, hospital admissions
* The Atrial Fibrillation Effect on QualiTy-of-Life Questionnaire (AFEQT) quality of life assessment AAD use: Class I/III AAD use will be permitted during the first two months post-ablation, during the post-procedure blanking period. At 2 month visit, AADs will be stopped in all patients. After the 2-month blanking period, AAD use will represent a treatment failure.

Cardioversions: Electrical/chemical cardioversions may be performed during the 2 month blanking period. If a subject is in AF near the completion of the blanking period at 2 months, a cardioversion should be performed so that the patient "exits" the Blanking period in sinus rhythm. After the 2-month blanking period, cardioversion will represent a treatment failure.

Early Exit: Any subject may cross over at 6 months. Early cross-over is allowed only in subjects with documented recurrence of AF/AT/AFL, plus one of the following:

1. AFEQT score at or below their baseline score for 3 consecutive months post-randomization may cross over, or
2. Subjects who have a drop in the AFEQT score of 10 or more points may cross over after 1 month

The treating cardiologist in follow-up, who is blinded to treatment assignment, will assess the persistence/worsening of symptoms and contact the core lab to confirm that AF/AT/AFL has recurred. After this confirmation, ablation will then be scheduled.

At the point of decision to cross-over / redo ablation, the patient will again take the AFEQT, HADS and Blinding questionnaire (this will serve in lieu of the 6 month assessments). Cross-over patients will be scheduled for PVI using pulsed-field ablation technology in the same manner as in the active ablation group. Beta-blockers and Ca-channel blockers will be preferentially used for symptom relief until the procedure.

Blinding

* Investigators: The operating physicians (electrophysiologists and anesthetists) will not be blinded to treatment assignment. As much as possible, site based study personnel who perform follow-up evaluations will remain blinded to subject treatment assignment.
* Subjects: Study personnel will be trained to avoid disclosing treatment status to study subjects. Study subjects will sign an informed consent that states that they will not be informed of their treatment status until the conclusion of their participation in the study.
* Core lab: The core lab, which will analyze ILR data, will remain blinded as much as possible consistent with accurate adjudication.
* Data and Safety Monitoring Board (DSMB): In general, the DSMB will review unblinded results in order to perform their function of protecting the integrity of the study and the rights, safety and welfare of study subjects.

Subjects will undergo a blinding assessment on day 1 post procedure, and at the 2 and 6 month visits. They will be asked whether they think they were assigned to the ablation group, the control group, or if they do not know. They will be asked to rate their degree of confidence in their answer on a scale of 1 to 5, with 5 pertaining to certainty.

ENDPOINTS

There will be two co-primary endpoints (assessed at six months):

1. Freedom from recurrent AF/AT/AFL (post two month blanking period): assessed as time to first recurrence (or to cross-over for Early Exits);
2. Quality of life according to the Atrial Fibrillation Effect on QualiTy of life (AFEQT) score at six months post ablation (or at cross-over for Early Exits).

Secondary endpoints

1. 6-month differences in AF/AT/AFL burden;
2. 6-month difference in HADS scores;
3. 12-month Freedom from recurrent AF/AT/AFL (post two month blanking period);
4. 12-month AFEQT scores (between treatment and control groups);
5. Correlation of AFEQT score with AF recurrence/burden data;
6. Unplanned Cardiovascular Hospitalization;
7. Procedure-related Major Complications;
8. Time to exit from assigned treatment.

AF/AFL/AT: episode of the corresponding arrhythmia that is recorded for review, where the recording contains at least 30 seconds of continuous interpretable signal.

ADVERSE EVENTS In both the control and treatment groups, the risks of sheath insertion in the femoral vein include access site complications (e.g., hematoma, fistula, pseudo-aneurysm, laceration, bleeding) potentially requiring surgical intervention. Risks of anesthesia in both groups include aspiration pneumonia, allergic reaction to medication, and cardiac arrhythmia.

In the treatment group, risks of catheter ablation include the following:

* Air embolism
* Anemia
* Cardiac tamponade or perforation
* Cardiac arrest or cardiac failure
* Cardiogenic shock
* Catheter entrapment potentially requiring endovascular or surgical intervention
* Conduction system injury, either transient or permanent, potentially requiring pacemaker insertion
* Coronary artery or vein injury
* Death
* Esophageal injury, ulcer or fistula
* Hemopericardium
* Hemoperitoneum
* Hemothorax
* Myocardial infarction / ischemia
* Nerve damage
* Pericardial effusion
* Pericarditis w
* Phrenic nerve injury with potential paralysis of the diaphragm and breathing impairment
* Pneumothorax
* PV injury, perforation or stenosis
* Stroke / transient ischemic attack

All safety analyses will utilize the adjudicated rather than site determination of an AE's characteristics in those instances where the CEC has adjudicated that characteristic to be different than the site's determination.

STATISTICAL RATIONALE AND STATISTICAL METHODS Originally, standard, frequentist approach with null hypothesis and significance testing was planned. However, during the study course, SHAM-PVI study was published showing the superiority of cryoablation over sham procedure, mostly in persistent AF patients). As such, to be able to enrol the minimum patient needed also for ethical reasons, the statistical approach was changed to Bayesian.

Bayesian statistics enables to adaptively adjust the sample size and compare it to previously published data. The Bayesian approach allows for continuous updates of treatment efficacy estimates based on newly acquired data. Moreover, Bayesian designs are increasingly being used not only in the early phases of clinical trials but are also gaining popularity in confirmatory trial phases. Bayesian adaptive designs thus enable continuous data monitoring without the need for additional adjustments for repeated testing. By using an Adaptive Bayesian design, we can calculate the predictive probability of success and decide whether to continue patient enrolment, terminate it due to achieved success, or end the study due to futility. Precisely because of more efficient resource utilization, shortening the duration of the study, and making more ethically responsible decisions since it reduces the number of patients exposed to less effective or placebo procedures, we preferred this method of adaptive Bayesian design in this study. Bayesian analysis thus provides not only flexibility and efficiency but also more credible and contextually informed statistical conclusions, which is key for accurately evaluating the true efficacy of catheter ablation compared to the SHAM group in this study. The use of Bayesian methods also allows for a direct and intuitive probabilistic interpretation of results.

For the AF recurrence primary endpoint, and with regard to the initial statistical plan, in the recently published EARLY-AF trial comparing cryoablation vs AADs, in which the effect of ablation was monitored using ILRs, one-year AF-freedom was present in 57.1% of ablated patients. In a recent study comparing PFA and radiofrequency ablation, one-year AF freedom (monitored using 24-hours Holter monitoring and weekly ECG transmissions) was achieved in 73% of patients in the PFA group. In the active-PFA treatment arm, 65% AF freedom at 6 month is a very conservative expectation in paroxysmal and persistent patients.

In eight studies comparing AADs with placebo using mixed monitoring methods (but no study used ILRs) with 655 patients, the success in placebo arms was 24.9% (95% CI 15-34). However, as noted, no study used ILR for monitoring, but no study experienced sham-procedure placebo that could be more effective than pharmacological placebo. For the AF Recurrence Primary Endpoint, in the sham-procedure arm, a maximum of 25% freedom at 6 months from AF could be maximally expected (and, as noted above, 65% in the active PFA arm). With β=80% and α=0.025, a total of 25 patients are required in each group, or 50 patients total. Due to potential crossover (outside the protocol), 60 patients would be required.

For the QoL Primary Endpoint, means are compared in independent samples, with the test of equality of means carried out at a 2-sided 0.05 level of significance, with a probability of 90% of rejecting the null hypothesis of equal proportions if the alternative holds. Assuming an AFEQT score of 50 in the Control group (with a S.D. of 20), and improvement to 70 in the Ablation group, a total of 25 patients are required in each group, or 50 patients total. Assuming the crossover (outside the protocol), 60 patients would be required. And finally, assuming minimal loss to follow-up, a total of 60 patients (30 per arm) will be enrolled. We will use a multiple hierarchical testing strategy where differences in AFEQT scores will be evaluated only if the test for time to AF/AT/AFL is statistically significant.

Formal rules for study termination The first (interim) analysis of a Bayesian adaptive study design will be done when the first 30 patients finish the 6 month follow-up. Then, subsequent statistical analyses will be done after each additional 10 patients finish 6 month follow-up. At each enrolment milestone, the Bayesian predictive probability that the trial will eventually demonstrate superiority for both co-primary endpoints is calculated. The study will be stopped if the Bayesian predictive probability of success is high for both co-primary endpoints when the current sample has been followed to 6 months (based on non-informative prior distribution), or for safety concerns. In particular, the study will be stopped if the posterior probability for the first (binary) co-primary endpoint (AF freedom) > 0.999, and for the second (continuous) co-primary endpoint (QoL) reaches extremely high probability of success (the Bayes Factor is > 100, indicating extreme evidence). Regarding safety rules, the entire study will be stopped if >5% patients in the sham group experience any adverse event including hospitalizations for AF recurrence.

On the other hand, enrolment stops for futility if the probability of ultimate success is low for both co-primary endpoints and the planned number of patients (n=60) finished the planned follow-up of 6 months.

Secondary Endpoint of Psychological Distress: As a secondary endpoint, we have planned for sufficient sample size to assess differences in psychological distress at 6 months between groups (using the Hospital Anxiety and Depression score, HADS). Based on the recently-published REMEDIAL study, where the mean baseline HADS score was approximately 12.3, we expect a mean baseline HADS score of 13 in our study since we are enriching for a more symptomatic cohort. We expect a mean HADS score at 6 months post-procedure to be 13 (with S.D. of 6; consistent with that observed in the REMEDIAL study) in the control group and 8 in the treatment group (an improvement by 5 points was observed with ablation in the REMEDIAL study). With β=80% and α=0.025, a total of 28 patients are required in each group, or 56 patients total.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years;
2. Paroxysmal or Persistent Atrial Fibrillation (but not long-standing Persistent AF);
3. AFEQT score ≤ 50.

Exclusion Criteria:

1. Any prior AF ablation procedure (or left atrial ablation procedure)
2. Untreated other arrhythmias (e.g. atrial flutter, SVT, VT, frequent PVCs);
3. Long-standing Persistent AF episodes (any continuous episodes lasting > 1 year);
4. Permanent AF;
5. No ECG evidence of AF episode >30 seconds in the 6 months prior to randomization;
6. LA size > 55 mm;
7. Hypertrophic cardiomyopathy;
8. Valve disease (any aortic stenosis, moderate or severe mitral regurgitation);
9. Left ventricular ejection fraction ≤ 35% according to echocardiogram within 6 months of randomization;
10. Moderate or severe pulmonary hypertension;
11. History of tachycardia-induced cardiomyopathy;
12. Symptomatic coronary artery disease;
13. Pregnancy;
14. Presence of an artificial valve;
15. Life expectancy less than two years;
16. Known medical condition or contraindication causing potential complications for interventional procedures or follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
AF freedom | 6 months
  Freedom from recurrent AF/AT/AFL (post two month blanking period): assessed as time to first recurrence (or to cross-over)
Quality of life | 6 months
  Quality of life according to the Atrial Fibrillation Effect on QualiTy of life (AFEQT) score at six months post ablation (or at cross-over for Early Exits) AFEQT is a 20-item questionnaire that asks about the degree to which different AF-related symptoms, treatment effects, and satisfaction with treatment have affected the patient over the past 4 weeks. The range is from 0 to 100. Lower scores indicate higher AF severity.

SECONDARY OUTCOMES:
AF burden | 6 months
  AF burden (percentage of time spent in AF) assessed using ILR.
Hospital Anxiety and Depression Score | 6 months
  Differences in Hospital Anxiety and Depression Score (HADS) between baseline (before randomization) and at 6 months Hospital Anxiety and Depression score, HADS, is a 14-item questionnaire assessing psychological distress. The range is from 0 to 42, or 0-21 for the assessment of Anxiety and 0-21 for assessment of Depression. The higher the score is, the higher level of Anxiety/Depression is present.
12-month Freedom from recurrent AF | 12 months
  Freedom from atrial fibrillation and regular atrial arrhythmias using implantable ECG loop recorder
12-month differences in quality of life | 12 months
  Quality of life assessed using AFEQT (Atrial Fibrillation Effect on QualiTy of Life ) questionnaire, range 1-20 AFEQT is a 20-item questionnaire that asks about the degree to which different AF-related symptoms, treatment effects, and satisfaction with treatment have affected the patient over the past 4 weeks. The range is from 0 to 100. Lower scores indicate higher AF severity.
Unplanned Cardiovascular Hospitalization | 12 month
  All hospitalizations for cardiovascular reason within 12 months. Only hospitalizations fo cardiovascular reason during 12 months will be evaluated, it means ofr myocardial infarcton, heart failure, thromboembolic events, and arrhythmias.
Procedure-related Major Complications | 2 months
  All adverse events associated with the procedure All complications that will be asigned to the procedure within the first one month after procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocenter, University Hospital Kralovske Vinohrady, Prague, Czechia